CLINICAL TRIAL: NCT02701101
Title: Evaluation of the SEM Scanner 200 for the Detection of Early Pressure Ulcers: A Multi-Site Longitudinal Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bruin Biometrics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Other
Other Study IDs: SEM200-008
Record Dates: First submitted 2016-02-11; First posted 2016-03-08 (Estimated); Results first posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Pressure Ulcers
Keywords: subepidermal moisture
MeSH Terms: conditions — Pressure Ulcer | interventions — Restraint, Physical

STUDY DESIGN:
Intervention Model Description: Enrolled subjects were evaluated once daily throughout the observation period for a minimum of 6 days to a maximum of 21 days upon enrollment or earlier exit from the study. Daily assessments were performed at the sacrum and both heels unless anatomical location(s) were not assessable. As it was unethical to withhold "standard of care" preventive measures from the enrolled subjects, in addition to the daily data collection of those listed above, daily prevention/intervention measures data was also collected. Prevention/intervention measures implemented may allow the physiology of the tissue to return to normal when intervened upon early in the pressure ulcer development pathway. Daily assessments included: 1. Risk Assessment (standard of care; Braden, Waterlow, or Norton) 2. Skin Assessment (Standard of Care visual skin assessments utilizing tactile and visual cues; and, 3. SEM Scanner readings ("test" variable in this study).
Who Masked: Care Provider, Outcomes Assessor
Masking Description: It was essential that both assessing teams' results were blinded to each other. Blinding between the "Specialist" and the "Generalist" teams was successfully upheld in this study. Data entry was structured in a manner restricting access based on roles and responsibilities defined in the study. The Study Investigators and Study Coordinators ("gate-keeper") were also diligent about ensuring blinding between the two assessing teams. The Principal Investigator or designated Co-Investigator were unblinded to the results of each study subject at the time of eCRF approval or exit for that subject. Prior to interim analysis, BBI's management team were also restricted to access the study's database, and thus were blinded to daily results. This further assures that no bias is introduced by the study sponsor to data collection.
Oversight: Data Monitoring Committee: No

ARMS (1):
- Daily Skin Assessments (SoC and SEM Scanner Readings) (Other): The SEM Scanner 200 measures sub-epidermal moisture ("SEM"), which has been studied as an indicator of localized edema characteristic of pressure-induced tissue damage. Daily assessments were performed at the sacrum and both heels unless the anatomical location(s) were not assessable. Daily assessments included:
  1. Risk Assessment (standard of care; Braden, Waterlow, or Norton)
  2. Skin Assessment (standard of care visual skin assessments utilizing tactile and visual cues)
  3. SEM Scanner readings ("test" variable in this study). Standard of care evaluations were conducted by individuals meeting the definition of Specialist specified in the study protocol whereas separate individuals meeting the definition of Generalist performed SEM Scanner 200 measurements. Specialists were blinded to the assessment by the Generalists, and vice versa.
  Interventions: Device: Use of SEM200 Scanner daily; Other: Assessment and treatment of Pressure Ulcers using SOC

INTERVENTIONS:
Device: Use of SEM200 Scanner daily — From enrollment to exit,daily SEM Scanner readings collected on Sacrum and Heels
Other: Assessment and treatment of Pressure Ulcers using SOC — Nurse review of Skin risk and skin assessment, notes in chart to assess the frequency to turn patient, use of a specialist bed to prevent or treat early pressure ulcers

SUMMARY:
This is a multi-site, longitudinal study to evaluate the use of the SEM Scanner as an adjunct to clinical judgment for detection of early pressure ulcers in patients before clinical judgment using signs of pressure ulcers from skin assessments. longitudinal study to evaluate the use of the SEM Scanner as an adjunct to clinical judgment for detection of early pressure ulcers in patients before skin assessments.

DETAILED DESCRIPTION:
All subjects are followed for a minimum of 6 days to a maximum of 21 days upon enrollment or until exit from the study . Enrolled subjects are assessed once daily throughout the follow-up period. Assessments are performed at the sacrum and both heels; if one or more locations are not assessable with the SEM Scanner, only the assessable locations are assessed. Each study site may include one or two wound care specialist (or a similarly trained clinician; the "Specialist") and one or two clinician/patient care provider(s) (the "Generalist") who perform assessments in the study.

Study assessments include (i) daily Risk Assessment and (ii) daily Skin Assessment performed by the Specialist blinded to the SEM readings; and (iii) daily SEM Scanner readings collected by the Generalist blinded to the Risk and Skin assessments. The outcome of interest is the diagnosis of a pressure ulcer by the Specialist using clinical judgment. The Specialist stages any diagnosed pressure ulcers according to NPUAP/EPUAP 2014 guidelines.

Note: If applicable, enrolled subjects continue to receive facility's standard of care practices for pressure ulcer preventive care. Participation in the study does not alter patient's standard of care.

This study involved two study objectives -

1. A primary objective to demonstrate the sensitivity and specificity of the SEM Scanner 200 in detecting early pressure ulcers before clinical judgment ("diagnose PU before clinical judgment").
2. A secondary objective to determine how early the SEM Scanner can detect signs before visually identified via clinical judgment ("time to detection").

ELIGIBILITY:
Inclusion Criteria:

1. Greater or equal to 55 years of age
2. At risk of developing a pressure ulcer at time of enrollment as defined by one or more of the following:

   1. PU Risk Score - Braden < 15; Waterlow ≥ 10; or Norton ≤ 18
   2. Poor mobility; e.g., Braden mobility subscore ≤ 2; Waterlow mobility subscore > 2; Norton mobility subscore ≤ 2; or poor mobility according to clinical judgment (chair- or bed-bound)
   3. Poor nutrition; e.g., Braden nutrition subscore ≤ 2; Waterlow nutrition subscore > 2; or poor nutrition according to clinical judgment
   4. Medical procedure (e.g. surgery, x-ray, etc.) involving immobility and inability to change position lasting 4 hours or longer
3. Evaluable by the study team for a minimum of 6 consecutive days upon enrollment
4. Willing and able to provide informed consent (or by proxy)

Exclusion Criteria:

1. Unhealed (including newly diagnosed) pressure ulcer at any anatomical site at the time of enrollment
2. Broken skin at the sacrum and both heels that prevents collection of SEM Scanner readings from all three anatomical locations; possible assessment at only one or two locations is not grounds for exclusion
3. Moisture lesion or incontinence associated dermatitis at the sacrum
4. Physical, structural, or other limitations preventing assessments required in this study (e.g., suspected or actual injury preventing turning)
5. Presence of any condition(s) or injury(ies) which compromises the subject's ability to complete this study
6. Per clinical decision of the study Investigator, diminished decision-making capacity which might impact compliance or completion with study procedures
7. Patient modesty concerns on the part of the subject (or their proxy) that might impact collection of SEM Scanner readings at the anatomical location (heels and sacrum) to be assessed

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2016-04; Primary Completion 2016-11 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Okonkwo H, Bryant R, Milne J, Molyneaux D, Sanders J, Cunningham G, Brangman S, Eardley W, Chan GK, Mayer B, Waldo M, Ju B. A blinded clinical study using a subepidermal moisture biocapacitance measurement device for early detection of pressure injuries. Wound Repair Regen. 2020 May;28(3):364-374. doi: 10.1111/wrr.12790. Epub 2020 Jan 21. PMID 31965682

RESULTS

PARTICIPANT FLOW:
Groups:
- Daily Skin Assessments (Standard of Care and SEM Readings): The SEM Scanner 200 measures sub-epidermal moisture ("SEM"), which has been studied as an indicator of localized edema characteristic of pressure-induced tissue damage. Daily assessments were performed at the sacrum and both heels unless the anatomical location(s) were not assessable. Daily assessments included:
  1. Risk Assessment (standard of care; Braden, Waterlow, or Norton)
  2. Skin Assessment (standard of care visual skin assessments utilizing tactile and visual cues)
  3. SEM Scanner readings ("test" variable in this study). Standard of care evaluations were conducted by individuals meeting the definition of Specialist specified in the study protocol whereas separate individuals meeting the definition of Generalist performed SEM Scanner 200 measurements. Specialists were blinded to the assessment by the Generalists, and vice versa.
  Use of SEM200 Scanner daily: From enrollment to exit,daily SEM Scanner readings collected on Sacrum and Heels
Period: Overall Study
Arm/Group | Daily Skin Assessments (Standard of Care and SEM Readings)
Started | 189
Completed | 189
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 189 subjects were enrolled but 7 subjects data were excluded from ITT analysis; non-analyzable data as per "valid Series" in the Statistical Analysis plan; three days of SEM scanner measurements with no more than one day missing between the three days of measurements and comprising no more than four observation days of SEM Scanner measurements.
Groups:
- Daily Skin Assessments (SoC and SEM Scanner Readings): The SEM Scanner 200 measures sub-epidermal moisture ("SEM"), which has been studied as an indicator of localized edema characteristic of pressure-induced tissue damage. Daily assessments were performed at the sacrum and both heels unless the anatomical location(s) were not assessable. Daily assessments included:
  1. Risk Assessment (standard of care; Braden, Waterlow, or Norton)
  2. Skin Assessment (standard of care visual skin assessments utilizing tactile and visual cues)
  3. SEM Scanner readings ("test" variable in this study). Standard of care evaluations were conducted by individuals meeting the definition of Specialist specified in the study protocol whereas separate individuals meeting the definition of Generalist performed SEM Scanner 200 measurements. Specialists were blinded to the assessment by the Generalists, and vice versa
  Use of SEM200 Scanner daily: From enrollment to exit,daily SEM Scanner readings collected on Sacrum and Heels
  Assessment and treatment o
Arm/Group | Daily Skin Assessments (SoC and SEM Scanner Readings)
Number analyzed (Participants) | 182
Age, Customized [Count of Participants; unit: Participants] — Greater than or equal to 55 years of age
  Participants
    >55 years of age | 182
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97
  Male | 85
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 158
  Unknown or Not Reported | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 44
  Native Hawaiian or Other Pacific Islander | 2
  Black or African American | 8
  White | 121
  More than one race | 4
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: The Sensitivity of the SEM Scanner Device (70% or Above) for Detecting Early Pressure Ulcers Before Routine Skin Assessments
Description: This study was powered to detect at least 70% sensitivity and 55% specificity of the device compared to the reference standard of clinical STA, with 95% confidence. A total of 189 patients were enrolled, of which 96.3% (n = 182) patients were listed as intent-to-treat (ITT).
Time Frame: A subject was included in the analysis when they had at least one "valid series" within 5 days of visual skin assessment identification of a pressure ulcer (6-21 observation days), or study exit when no pressure ulcer was identified.
Measure: Number (95% Confidence Interval); unit: percentage of true positives
Arm/Group | Daily Skin Assessments (SoC and SEM Scanner Readings)
Number analyzed (Participants) | 182
percentage of true positives | 87.5 [74.8 to 95.3]

2. Primary Outcome: The Specificity of the SEM Scanner Device (60% or Above) for Detecting Early Pressure Ulcers
Description: The use of specificity as an end point was recognized, before study inception, as a worst-case assessment for the SEM test because it classes all results in which a pressure ulcer did not visibly manifest (STA negative) but where changes in SEM were observed (SEM positive) as false positive results.
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of True negatives
Arm/Group | Daily Skin Assessments (SoC and SEM Scanner Readings)
Number analyzed (Participants) | 182
Percentage of True negatives | 32.9 [28.3 to 37.8]

3. Secondary Outcome: Determine the Average Number of Days Between Detection of Early Pressure Ulcers Using the SEM Scanner and Diagnosis of Pressure Ulcers Through Clinical Judgement ("Time to Detection").
Description: The measure for secondary endpoint is the Number of Days between pressure ulcer diagnosis by clinical judgment of the Specialist and the first day of SEM Scanner delta >0.5 ("time to detection"). For the secondary endpoint, the first measurement of the Valid Series can be at any time during the subject's participation.
Time Frame: as for outcome 1
Population: Secondary endpoint is only analyzed for subjects identified with positive detection (pressure ulcer by Specialist and SEM Scanner with delta >0.5).The Number of Days is the difference between pressure ulcer diagnosis by clinical judgment of the Specialist and the first day of SEM Scanner delta >0.5 ("time to detection").
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Daily Skin Assessments (Standard of Care and SEM Readings)
Number analyzed (Participants) | 182
days | 4.74 (2.39)

ADVERSE EVENTS:
Time Frame: A subject was included in the analysis when they had at least one "valid series" within 5 days of visual skin assessment identification of a pressure ulcer (6-21 observation days), or study exit when no pressure ulcer was identified.
Description: All enrolled 189 subjects were scanned using the SEM scanner and Visual Skin Assessments. AE events could not be distinguished by arm. All SAE's (clinicaltrials.gov definition) and any device related AEs were defined as "SAEs" consistent with the non-significant risk classification/indication for the device. AEs (clinicaltrials.gov definition) and unrelated to the device were defined as AE's. SAE, AE events are reported in enrolled 189 subjects as opposed to ITT analysis for 182.
Arm/Group | Daily Skin Assessments (Standard of Care and SEM Readings)
All-Cause Mortality (participants affected / at risk) | 4/189
Serious Adverse Events (participants affected / at risk) | 0/189
Other Adverse Events (participants affected / at risk) | 1/189
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Daily Skin Assessments (Standard of Care and SEM Readings) (N=189)
Unrelated to device AE (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator and Institution shall be free to publish and present the results and data from the Study per the following conditions.The manuscript or abstract proposed to be published or presented shall be submitted to Sponsor for review and comment at least forty-five (45) days prior to submission for publication or presentation to allow Sponsor to protect its rights to any patentable inventions disclosed in such publication or presentation.